CLINICAL TRIAL: NCT04398004
Title: Anti-inflammatory Clarithromycin to Improve SARS-CoV-2 (COVID-19) Infection Early: The ACHIEVE Open-label Non-randomized Clinical Trial
Brief Title: Anti-inflammatory Clarithromycin for Improving COVID-19 Infection Early
Acronym: ACHIEVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ACHIEVE; 2020-001882-36 (EudraCT Number)
Record Dates: First submitted 2020-05-17; First posted 2020-05-21 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: COVID-19; Virus Diseases; Corona Virus Infection
Keywords: COVID-19; SARS-CoV-2; Clarithromycin; Hydroxychloroquine
MeSH Terms: conditions — COVID-19; Virus Diseases; Coronavirus Infections | interventions — Clarithromycin

STUDY DESIGN:
Intervention Model Description: Treatment with clarithromycin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clarithromycin arm (Experimental): Treatment will last for seven days. Every patient will receive one tablet of 500 mg of clarithromycin every 12 hours. It is explicitly stated that all other treatment is allowed with the only exclusion the parallel intake of a) any other drug of the macrolide class of antibiotics; and/or b) hydroxychloroquine or chloroquine phosphate. Drugs contraindicated with the intake of clarithromycin are also not allowed, as they are described in the local label information.
  Interventions: Drug: Clarithromycin

INTERVENTIONS:
Drug: Clarithromycin — Treatment with 500 mg Clarithromycin orally twice daily for seven days
  Other Names: Klaricid

SUMMARY:
Recent information appearing from different countries suggest that treatment of Coronavirus disease 2019 (COVID-19) with hydroxychloroquine or with a combination of hydroxychloroquine and azithromycin has either an indifferent effect on viral replication or substantial cardiotoxicity. This is a clinical trial aiming to prove that addition of oral clarithromycin to treatment regimen of COVID-19 is associated with early clinical improvement and attenuation of the high inflammatory burden of the host. The study will not comprise a placebo-comparator group since this is considered inappropriate in an era of a pandemic with substantial global mortality.

DETAILED DESCRIPTION:
Humanity is experiencing since December 2019 a new pandemic by the novel SARS Coronavirus-19 (SARS-CoV-2). As of March 25 2020 418,099 documented case were reported worldwide; 18,608 patients died. The analysis of the clinical characteristics of these patients showed that the natural course of this disease, known with the acronym COVID-19, is several times unpredictable. Most patients who develop pneumonia do not have worrying symptoms although their chest X-ray or chest computed tomography may be positive for diffuse infiltrates. Suddenly a certain proportion of these patients deteriorate into severe respiratory failure; this usually takes place between the 5th and the 10th day of illness and arrives without any preceding symptom. Published evidence suggests that this is due to the sudden arrival of an acute pro-inflammatory reaction of the host. With this in mind, it is reasonable to make the assumption than the early treatment with an agent that can efficiently modulate the host response and prevent sudden hyper-inflammatory reaction may prevent the development of severe respiratory failure (SRF).

The new guidelines published by the American Thoracic Society in 2019 clearly suggest that the management of community-acquired pneumonia (CAP) should rely on the combination of β-lactam antibiotics with macrolides. This position statement is pretty much influenced by the retrospective analyses of observational studies and of their meta-analyses in showing that the addition of a macrolide improves survival from severe CAP. Since patients leave in an era of antimicrobial resistance, it is profound that survival benefit is linked to the anti-inflammatory properties of the macrolide class of antibiotics. These properties are not only limited to the attenuation of the production of pro-inflammatory mediators but they involve the enhancement of pathogen clearance.

With this in mind, a small open-label trial among patients with COVID-19 showed better viral containment as assessed by the persistence of the virus in respiratory secretions, when patients were treated with a combination of azithromycin and hydroxychloroquine. However, the clinical benefit coming from this study has not yet been published. Contrary to azithromycin, clinical evidence suggests that clarithromycin is associated with substantial clinical benefit among critically ill patients. Two randomized clinical studies in a total of 800 patients with sepsis have shown 28-day survival benefit among the most severe cases. One of these studies enrolled patients with sepsis and ventilator-associated pneumonia; among 100 patients allocated to placebo treatment 40% survived until day 90; this was 57% among clarithromycin-treated patients.

In recent publication coming from the research network of the Hellenic Sepsis Study Group (HSSG) 130 patients with CAP were treated with a combination of β-lactam and clarithromycin. These patients were compared with 130 patients treated with a combination of β-lactam and azithromycin. Groups were well-matched for severity and comorbidities; 28-day mortality was 20.8% and 33.8% respectively.

Based on the above analysis, it seems likely that treatment of patients with COVID-19 with oral clarithromycin will substantially increase their anti-inflammatory properties and decrease the chances for development of severe respiratory failure.

As stated above, the efficacy of the treatment combination of hydroxychloroquine with azithromycin is based on results coming from only six patients. Since the publication of these data other, yet unpublished, reports have appeared in the internet challenging the treatment efficacy of this combination. These results show that treatment with hydroxychloroquine either single or in combination with azithromycin have either an indifferent effect on viral replication or even a deleterious effect on the patient due to cardiotoxicity. With this in mind it is obvious that macrolide treatment in COVID-19 patients many of which have coronary heart disease and chronic heart failure as comorbidities should be administered without hydroxychloroquine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Male of female gender
* Written informed consent provided by the patients or by a first-degree relative in case of patients unable to consent
* In case of women, unwillingness to remain pregnant during the study period achieved either by their partner using condom or by themselves using oral contraceptives.
* Confirmed infection by SARS-CoV-2 virus
* Infection of the upper respiratory tract or of the lower respiratory tract

Exclusion Criteria:

* Age below 18 years
* Denial of written informed consent
* Intake of any macrolide for the current episode of infection under study
* Intake of hydroxychloroquine or chloroquine phosphate.
* Presence of severe respiratory failure
* Oral or intravenous intake of corticosteroids defined as any more than 0.4mg/kg daily intake of equivalent prednisone for the last 15 days
* Neutropenia defined as an absolute neutrophil count below 1,000/mm3
* Presence of any contraindications for the study drugs as stated in local label information
* QTc interval at rest electrocardiogram ≥500 msec or history of known congenital long QT syndrome
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Clinical outcome negative for two parameters(hospital admission/disease progression) | Day 1 to Day 8
  This is defined on day 8 (End of Treatment - EOT). Patients with upper respiratory tract infection by SARS-CoV-2 meet the study primary endpoint if they were not admitted to hospital or their symptoms did not progress to lower respiratory tract infection.
  Patients who develop by day 8 severe respiratory failure do not meet the study primary endpoint.
At least 50% change of the score of respiratory symptoms from the baseline | Day 1 to Day 8
  This is defined on day 8 (EOT visit). Patients with lower respiratory tract infection by SARS-CoV-2 meet the primary endpoint if they present at least 50% decrease of the score of respiratory symptoms from the baseline. This score is the sum of scoring for the symptoms of cough, dyspnea, purulent sputum expectoration and pleuritic chest pain.
  Patients who develop by day 8 severe respiratory failure do not meet the study primary endpoint. Score ranges from 0 (no symptoms) to 9 (worst for all symptoms).

SECONDARY OUTCOMES:
Comparison of two parameters with historical comparators from Hellenic Sepsis Study Group Database | Day 1 to Day 8
  Evaluation of need of hospitalization, SARS-CoV-2 infection progression from upper to lower respiratory tract infection, between baseline and study visit day 8 will be compared with historical comparators from Hellenic Sepsis Study Group Database
Comparison of the score of respiratory symptoms with historical comparators from Hellenic Sepsis Study Group Database | Day 1 to Day 8
  Respiratory score between baseline and study visit day 8 will be compared with historical comparators from Hellenic Sepsis Study Group Database.
  This score is the sum of scoring for the symptoms of cough, dyspnea, purulent sputum expectoration and pleuritic chest pain.Score ranges from 0 (no symptoms) to 9 (worst for all symptoms).
Clinical outcome negative for two parameters(hospital admission/disease progression) on day 4 | Day 4
  Comparison of clinical data (need of hospitalization, the infection progression of SARS-CoV-2 from upper to lower respiratory tract infections) in enrolled patients between baseline and study visit day 4 Patients who develop by day 4 severe respiratory failure do not meet the study secondary endpoint.
At least 50% change of the score of respiratory symptoms from the baseline on day 4 | Day 4
  This is defined on day 4 (5th visit). Patients with lower respiratory tract infection by SARS-CoV-2 meet the secondary endpoint if they present at least 50% decrease of the score of respiratory symptoms from the baseline. This score is the sum of scoring for the symptoms of cough, dyspnea, purulent sputum expectoration and pleuritic chest pain.
  Patients who develop by day 4 severe respiratory failure do not meet the study secondary endpoint. Score ranges from 0 (no symptoms) to 9 (worst for all symptoms).
Range of development of severe respiratory failure | Day 1 to Day 14
  Evaluation of range of enrolled patients who develop severe respiratory failure between baseline and day 14 (TOC VISIT). Severe respiratory failure is defined by presence of all of the following
  * pO2/FiO2 less than 150
  * Need for mechanical or non-mechanical ventilation (CPAP)
Range of hospital readmission until day 14 | Day 1 to Day 14
  Evaluation of hospital readmission until day 14 (TOC VISIT) from enrollment defined as either need of re-hospitalization for discharged patients or any need for hospitalization of out-patients.
Change of viral load in respiratory secretions from baseline on day 8 | Day 1 to Day 8
  Comparison of Real Time - Polymerase Chain Reaction (RT-PCR) results for SARS-CoV-2 viral load in rhinopharyngeal samples of enrolled patients at days 1, 4 and 8
Change of function of monocytes at days 1 and 8 | Day 1 to Day 8
  Change of cytokine production of monocytes in enrolled patients with upper/lower respiratory tract infection at days 1 and 8 (EOT) visit; monocytes will be stimulated for 24 hours with SARS-CoV-2 purified antigens for the production of TNFα. This will be analyzed separately for patients with upper and with lower respiratory tract infection
Change of function of Th1 cells at days 1 and 8 | Day 1 to Day 8
  Change of cytokine production of Th1 cells in enrolled patients with upper/lower respiratory tract infection at days 1 and 8 (EOT) visit; Th1 cells will be stimulated for 24 hours with SARS-CoV-2 purified antigens for the production of IFNγ. This will be analyzed separately for patients with upper and with lower respiratory tract infection.
Change of function of Th2 cells at days 1 and 8 | Day 1 to Day 8
  Change of cytokine production of Th2 cells in enrolled patients with lower respiratory tract infection at days 1 and 8 (EOT) visit; Th2 cells will be stimulated for 24 hours with SARS-CoV-2 purified antigens for the production of IL6. This will be analyzed separately for patients with upper and with lower respiratory tract infection.
Change of serum interleukin-6 (IL-6) cytokine levels between days 1 and 8 | Day 1 to day 8
  Change of the serum levels of interleukin-6 (IL-6) of enrolled patients between day 1 and day 8 (EOT VISIT); this is also analyzed separately for patients with upper and with lower respiratory tract infection
Change of serum interleukin-8 (IL-8) cytokine levels between days 1 and 8 | Day 1 to day 8
  Change of the serum levels of interleukin-8 (IL-8) of enrolled patients between day 1 and day 8 (EOT VISIT); this is also analyzed separately for patients with upper and with lower respiratory tract infection
Change of serum human beta defensin-2 (hBD-2) between days 1 and 8 | Day 1 to day 8
  Change of the serum levels of human beta defensin-2 (hBD-2) of enrolled patients between day 1 and day 8 (EOT VISIT); this is also analyzed separately for patients with upper and with lower respiratory tract infection
Change of cytokine levels interleukin-6 (IL-6) at the rhinopharynx between days 1,4 and 8 | Day 1 to day 8
  Change of rhinopharynx levels of interleukin-6 (IL-6) of enrolled patients between day 1, day 4 and day8 (EOT visit); this is also analyzed separately for patients with upper and with lower respiratory tract infection
Change of interleukin-1 (IL-1) cytokine levels at the rhinopharynx between days 1,4 and 8 | Day 1 to day 8
  Change of rhinopharynx levels of interleukin-1 (IL-1) of enrolled patients between day 1, day 4 and day8 (EOT visit); this is also analyzed separately for patients with upper and with lower respiratory tract infection
Change of the IL-10/TNFα ratio between days 1 and 8 | Day 1 to Day 8
  Comparison of the Interleukin-10/Tumor Necrosis Factor α (IL-10/TNFα) ratio in enrolled patients at days 1 and 8; this is also analyzed separately for patients with upper and with lower respiratory tract infection

CONTACTS AND LOCATIONS:
Overall Officials: Garyfallia Poulakou, MD, PhD, Principal Investigator — National Kapodistrian University of Athens, Medical School
Locations (9):
- Greece (9):
  - COVID-19 Department, General Hospital of Attica SISMANOGLEIO-AMALIA FLEMING, Marousi, Athens
  - 2nd Department of Internal Medicine, General Hospital of Nikaia, Piraeus, Attica
  - 2nd Department of Internal Medicine, University General Hospital of Alexandroupolis, Alexandroupoli
  - 1st University Department of Internal Medicine, LAIKO General Hospital of Athens, Athens
  - 2nd University Department of Internal Medicine, IPPOKRATEION General Hospital of Athens, Athens
  - 3rd University Department of Internal Medicine, General Hospital of Chest Diseases of Athens I SOTIRIA, Athens
  - 1st Department of Internal Medicine, General University Hospital of Ioannina, Ioannina
  - 2nd Department of Internal Medicine, General Hospital of Piraeus "Tzaneio", Piraeus
  - 1st Department of Internal Medicine, AHEPA University General Hospital of Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsiakos K, Tsakiris A, Tsibris G, Voutsinas PM, Panagopoulos P, Kosmidou M, Petrakis V, Gravvani A, Gkavogianni T, Klouras E, Katrini K, Koufargyris P, Rapti I, Karageorgos A, Vrentzos E, Damoulari C, Zarkada V, Sidiropoulou C, Artemi S, Ioannidis A, Papapostolou A, Michelakis E, Georgiopoulou M, Myrodia DM, Tsiamalos P, Syrigos K, Chrysos G, Nitsotolis T, Milionis H, Poulakou G, Giamarellos-Bourboulis EJ. Early Start of Oral Clarithromycin Is Associated with Better Outcome in COVID-19 of Moderate Severity: The ACHIEVE Open-Label Single-Arm Trial. Infect Dis Ther. 2021 Dec;10(4):2333-2351. doi: 10.1007/s40121-021-00505-8. Epub 2021 Aug 6. PMID 34363189